CLINICAL TRIAL: NCT01189305
Title: Behavioral Couples Therapy for Female Drug-Abusing Patients
Acronym: CPW-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Timothy J. O'Farrell, Professor of Psychology, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA025618 (NIH); 1R01DA025618 (NIH)
Record Dates: First submitted 2010-08-16; First posted 2010-08-26 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Drug Abuse
Keywords: Drug Abuse; Female Patients
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Couples Therapy (Experimental)
  Interventions: Behavioral: Behavioral Couples Therapy
- Individual Drug Counseling (Experimental)
  Interventions: Behavioral: Individual Drug Counseling

INTERVENTIONS:
Behavioral: Behavioral Couples Therapy — Behavioral Couples Therapy
  Arms: Behavioral Couples Therapy
Behavioral: Individual Drug Counseling — Individual Drug Counseling
  Arms: Individual Drug Counseling

SUMMARY:
In treating drug addiction, many studies of male patients show Behavioral Couples Therapy (BCT) helps the whole family (the drug abuser, the relationship partner, and their children) and is more effective than typical individual and group counseling. Only one study of BCT has been done with female drug-abusing patients, and results were promising but not definitive. The proposed study will test with married or cohabiting female drug-abusing patients whether BCT will produce more positive outcomes for the women, their male partners, and their children than standard individual counseling for the patient alone.

ELIGIBILITY:
Inclusion Criteria:

* female patients with primary drug abuse diagnosis & their relationship partners
* patient married or cohabiting with relationship partner
* partner without current alcohol or drug problem

Exclusion Criteria:

* both patient and partner without severe mental health disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2009-07; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
percent days abstinent from illicit drugs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J O'Farrell, PhD, Principal Investigator — Harvard University
Locations (1):
- AdCare Hospital of Worcester Inc., Worcester, Massachusetts, United States